CLINICAL TRIAL: NCT03285906
Title: An Exploratory Clinical Study of Apatinib for the 2nd Treatment of Esophageal Cancer or Esophageal and Gastric
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AHEAD-HBE001
Record Dates: First submitted 2017-08-21; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-07

CONDITIONS: Esophagus Cancer, Stage III; Esophageal Gastric Cardia Type Metaplasia; Esophagus Cancer, Stage IV
MeSH Terms: conditions — Esophageal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Apatinib：500 mg，po，qd
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Targeted therapy Apatinib：500 mg，po，qd
  Other Names: YN968D1

SUMMARY:
The purpose of this Phase II, Open-label, single arm, exploratory study is to evaluate the efficacy and the safety of Apatinib（500mg/d）for the second - line treatment of esophageal cancer or esophageal and gastric

DETAILED DESCRIPTION:
This study is a prospective,single-center,single arm,Ⅱ exploratory study.To explore the clinical study of the efficacy and safety of the treatment of vegfr-2 high expression by apatinib mesilate.The main research object for first-line treatment failure Ⅲ/Ⅳ integration of a period of esophageal or gastric esophagus cancer patients.The main purpose of the study was to evaluate apatinib for the median PFS of the esophageal and esophageal gastric junction carcinoma of the esophagus with high expression of VEGFR-2. The objective of secondary research is to evaluate the safety of apatinib for second-line treatment of esophageal and esophageal gastric junction cancer Objective Response Rate (CR + PR) and median OS and explore the relationship between VEGFR-2 high expression and apatinib efficacy and related prognostic factors. Thirty patients were enrolled in the study group. The group was expected to be enrolled in the group for 24 months, followed by 6 months of follow-up and 6 months of data statistics. The drug regimen was a single drug apatinib 500mg qd Po.Please refer to the CRF table for details.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 75 years of age
* Have failed for 1 lines of chemotherapy
* ECOG performance scale 0 - 2.
* Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥ 90g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.25×the upper limit of normal(ULN), and serum transaminase≤2.5×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.5 x ULN, creatinine clearance rate ≥ 50ml/min.
* Life expectancy of more than 12 months

Exclusion Criteria:

* Existing therapy related toxicity of prior chemotherapy and/or radiation therapy
* Intercurrence with one of the following: hypertension, coronary artery disease, arrhythmia and heart failure
* Any factors that influence the usage of oral administration
* The center of the tumor invaded local large blood vessels
* Within 4 weeks before the first use of drugs, occurs pulmonary hemorrhage (≥ CTCAE class 2) or other parts' hemorrhage (≥ CTCAE class 3).
* Within 6 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc.
* Less than 4 weeks from the last clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Through study completion, an average of 1 year
  No progress in survival (PFS) is to use the RECIST 1.1 standard to assess the progress of the evaluation of the population without progress.The date of the first occurrence of a disease or any cause of death from a random date to the first occurrence.

SECONDARY OUTCOMES:
Objective Response Rate | Through study completion, an average of 0.5 year
  Objective Response Rate(ORR):The proportion of patients who have been reduced to a certain amount and maintained a certain amount of time, including the CR + PR case.
median Overall Survival | Through study completion, an average of 1.5 year
  median Overall Survival (mOS):It means that 50% of patients start from randomization to the time of death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Pan Zhanyu, Master, Principal Investigator — 86-13752570372
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
PFS data of patients in this trial are expected to be Shared